CLINICAL TRIAL: NCT03550937
Title: Hospital-based Surveillance of Severe Rotavirus Gastroenteritis and Diversity of Circulating Rotavirus Strains in Young Taiwanese Children
Brief Title: Hospital-based Surveillance of Rotavirus Gastroenteritis in Young Taiwanese Children
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201310064RINA
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Rotavirus Gastroenteritis, Young Taiwanese Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rotavirus remains among the leading causes of pediatric gastroenteritis requiring hospitalization in the world. Surveillance studies revealed that more than 90% of the global circulating rotavirus strains were predominated by several major genotypes. Clinical trials and post-marketing studies have demonstrated that the currently available rotavirus vaccine can provide sufficient protection against strains of the prevalent genotypes. However, the emerging strains with new genotypes were increasingly reported in the past decade, an ongoing surveillance of the strain changes is needed in the regions where the pediatric population is either fully or partly immunized. In this project, the investigators will setup a hospital-based gastroenteritis surveillance network by incorporating 8 major hospitals in northern, central, southern and eastern Taiwan. From 2013 to 2015, children aged 5 years or younger hospitalized to one of the 8 sentinel hospitals due to acute gastroenteritis will be screened for rotavirus infection, and viral proteins 7 [VP7] (G type) and viral proteins 4 [VP4] (P type) genotypes of rotavirus will be determined for each infected case. The demographics and clinical manifestations of study subjects will also be collected and analyzed. Through this project, the investigators will be able to detect emerging genotypes of rotavirus and delineate the strain distribution during the two years of study in Taiwan. The investigators can also have more comprehensive understanding of the epidemiology of rotavirus regarding to the incidence, disease characteristics, temporal and geographic variations of severe rotavirus gastroenteritis in Taiwanese children. Results from this project will provide valuable information for future implementation of mass immunization against rotavirus in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* aged less than 60 months,
* hospitalized in 1 of the 8 hospitals,
* having diarrhea not caused by any known underlying diseases.

Exclusion Criteria:

* No

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized children having diarrhea and less than 60 months of age
Sampling Method: Non-Probability Sample
Enrollment: 5040 (Actual)
Dates: Start 2013-12-11 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
monitor the strain diversity of rotavirus in Taiwan | 4 years
  monitor the strain diversity of rotavirus in Taiwan, including the individual serotype prevalence and emerging genotypes

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - Chang Bing Show Chwan Memorial Hospital, Chang-hua
  - Chang Hua Show Chwan Memorial Hospital, Chang-hua
  - National Taiwan University Hospital Yun-Lin Branch, Douliu
  - Buddhist Tzu Chi General Hospital, Hualien Tzu Chi Medical Center, Hualien City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Children's Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No